CLINICAL TRIAL: NCT06678178
Title: Testing Climate Impact Menu Labels Influence on Nutrition Quality of Fast-Food Selections: A Pilot Study
Brief Title: Climate Impact Label Design and Fast-Food Meal Selection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of California, Davis (Other); Harvard School of Public Health (HSPH) (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00030419; 1R01DK139327-01 (NIH); IRB00030419 (Other: Johns Hopkins Bloomberg School of Public Health IRB)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Food Selection
Keywords: food labeling; climate labeling; choice behavior
MeSH Terms: conditions — Food Preferences | interventions — Product Labeling

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to view a fast-food menu with one of five labeling schemes applied: (1) a QR code on all items (control); (2) a high climate impact warning label on high impact items; (3) traffic light labeling on all items by level of impact; (4) climate grade labels on all items by level of impact; and (5) numeric labels on all items. All fast-food menus will include main items, sides, desserts, and drinks. Labels will only appear alongside main menu items and will be assigned using thresholds for greenhouse gas emissions set a priori in kilograms of CO2 equivalent per kilogram of food. Participants will be instructed to select a hypothetical lunch meal order. The investigators will record participant meal selections and, using publicly available nutritional information for each item selected, calculate a score of overall meal healthfulness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Control (QR) Labels (Placebo Comparator): A black label featuring a QR code and white text that reads "SCAN HERE" will be placed beneath all main menu items. Explanatory text describing the label's meaning will be displayed at the top of the menu.
  Interventions: Behavioral: Control (QR) Labels
- Warning High Climate Impact Labels (Experimental): A red icon-plus-text label that reads "WARNING: HIGH CLIMATE IMPACT" in white text will be placed beneath main menu items with a high climate impact using a predetermined threshold of estimated greenhouse gas emissions set at >=9.2 kgCO2e. Labels will include a white globe icon directly preceding the label text. Explanatory text describing the label's meaning will be displayed at the top of the menu.
  Interventions: Behavioral: Warning High Climate Impact Labels
- Traffic Light Labels (Experimental): Traffic Light labels will be placed beneath all main menu items. Using predetermined estimated greenhouse gas emission thresholds, each item will be assigned one of three icon-plus-text labels within this scheme: low-, medium-, or high-impact label, set in kgCO2e at <2.6, >=2.6 & <9.2, and >=9.2, respectively. Each will read, "HIGH CLIMATE IMPACT" within a red label, "MED. CLIMATE IMPACT" in a yellow label, and "LOW CLIMATE IMPACT" in a green label. Text for all labels written in white, and a white globe icon will precede the text. Explanatory text describing the meaning of the labels will be displayed at the top of the menu.
  Interventions: Behavioral: Traffic Light Labels
- Climate Grade Labels (Experimental): Climate Grade labels will be placed beneath all main menu items, using predetermined estimated greenhouse gas emission thresholds to assign one of five icon-plus-text labels which indicate a specific climate impact grade (A, B, C, D, and F). Thresholds are set in kgCO2e as follows: [A] <1.7, [B] >=1.7 & <2.6, [C] >=2.6 & <9.2, [D] >=9.2 & <28, [F] >=28. All labels are solid black with a white globe icon followed by white text which reads "CLIMATE GRADE". On the left side of each label, a grade is displayed, capitalized and in a white font within a solid-colored box. The color of the box corresponds with each letter grade: A = dark green, B = light green, C = yellow, D = orange, F = red. Beneath the letter grade, a gradient of all possible grades is displayed horizontally in smaller font, each grade atop a small solid box in the respective grade color. Explanatory text describing the meaning of the labels will be displayed at the top of the menu.
  Interventions: Behavioral: Climate Grade Labels
- Numeric Carbon Footprint Labels (Experimental): Numeric Carbon Footprint labels will be placed beneath all main menu items and display the estimated greenhouse gas emissions in kilograms of carbon dioxide equivalents (kgCO2e) for each item. All labels have a solid black background and an icon-plus-text design. A white globe icon is followed by text stating the value of the items estimated emissions and the unit "kgCO2e". Explanatory text describing the meaning of the labels will be displayed at the top of the menu.
  Interventions: Behavioral: Numeric Carbon Footprint Labels

INTERVENTIONS:
Behavioral: Control (QR) Labels — Participants will view a fast-food restaurant menu including main, side, dessert, and drink items. Each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Control (QR) labels will be displayed beneath each item. Participants will be instructed to select up to 4 menu items for a hypothetical meal order.
  Arms: Control (QR) Labels
Behavioral: Warning High Climate Impact Labels — Participants will view a fast-food restaurant menu including main, side, dessert, and drink items. Each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Warning High Climate Impact labels will be displayed beneath select items. Participants will be instructed to select up to 4 menu items for a hypothetical meal order.
  Arms: Warning High Climate Impact Labels
Behavioral: Traffic Light Labels — Participants will view a fast-food restaurant menu including main, side, dessert, and drink items. Each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Traffic Light labels will be displayed beneath each item. Participants will be instructed to select up to 4 menu items for a hypothetical meal order.
  Arms: Traffic Light Labels
Behavioral: Climate Grade Labels — Participants will view a fast-food restaurant menu including main, side, dessert, and drink items. Each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Climate Grade labels will be displayed beneath each item. Participants will be instructed to select up to 4 menu items for a hypothetical meal order.
  Arms: Climate Grade Labels
Behavioral: Numeric Carbon Footprint Labels — Participants will view a fast-food restaurant menu including main, side, dessert, and drink items. Each menu item will be displayed with an image of the item, name, price, and total calories. For main items only, Numeric Carbon Footprint labels will be displayed beneath each item. Participants will be instructed to select up to 4 menu items for a hypothetical meal order.
  Arms: Numeric Carbon Footprint Labels

SUMMARY:
The primary objective of this study is to test the relative effects of climate-impact menu label designs on the healthfulness of consumers' fast-food meal choices. Participants will complete a hypothetical online meal ordering task using a survey which emulates the online menu of a burger restaurant chain. Participants will be randomized for exposure to menus featuring one of five labeling conditions. Secondary objectives include examining total greenhouse gas emissions per meal order and, through a post-order survey, perception of labels between the conditions.

DETAILED DESCRIPTION:
This online randomized trial will test the relative effects of climate impact menu label designs on the healthfulness of consumers' fast-food meal choices and perceptions of menu items. The survey research firm CloudResearch will recruit a sample of 6,250 adults aged 18 years and older who speak English and reside in the United States.

Participants will complete a between-subjects online experiment in which the participants will be randomized to view a fast-food online ordering menu with one of five labeling schemes applied: (1) a QR code on all items (control); (2) a high climate impact warning label on high impact items; (3) traffic light labels on all items by level of impact; (4) climate grade labels on all items by level of impact; and (5) numeric carbon footprint labels on all items. All fast-food menus will include main items, sides, desserts, and drinks. Labels will only appear alongside main menu items and will be assigned using thresholds for greenhouse gas emissions set a priori in kilograms of carbon dioxide (CO2) equivalent per kilogram of food. Participants will be instructed to select up to 4 menu items for a hypothetical meal order. After completing the meal ordering task, participants will be prompted to answer questions about the perception of the labeling condition which the participants were randomized to view, perception of the relative effectiveness of all labels in this experiment, and personal values, dietary patterns, and other demographic information.

The primary outcome will be the healthfulness of meal orders selected from the online menu, indicated by a modified Nutrient Profile Index meal score for all food items ordered. Secondary outcomes will be total greenhouse gas emissions per meal ordered, total calories ordered, whether a sugar-sweetened beverage was ordered, and perceived message effectiveness of the climate-impact labels.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Member of the CloudResearch panel
* Residing in the United States

Exclusion Criteria:

* Under 18 years of age
* Not residing in the United States
* Completed the survey implausibly quick based on the distribution of the time to complete the survey among all participants
* Failed the built-in Qualtrics survey fraud detection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6622 (Actual)
Dates: Start 2024-12-02 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wolfson, PHD MPP, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
Started | 1320 | 1339 | 1332 | 1305 | 1326
Completed | 1245 | 1245 | 1257 | 1229 | 1245
Not Completed | 75 | 94 | 75 | 76 | 81

BASELINE CHARACTERISTICS:
Population: Participants who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels | Total
Number analyzed (Participants) | 1245 | 1245 | 1257 | 1229 | 1245 | 6221
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (17) | 47 (17) | 48 (17) | 46 (17) | 47 (17) | 47 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 629 | 633 | 670 | 658 | 643 | 3233
  Male | 616 | 612 | 587 | 571 | 602 | 2988
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 174 | 177 | 188 | 168 | 171 | 878
  Not Hispanic or Latino | 1071 | 1068 | 1069 | 1060 | 1074 | 5342
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 18 | 26 | 19 | 23 | 105
  Asian | 56 | 57 | 46 | 56 | 55 | 270
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 171 | 160 | 166 | 156 | 165 | 818
  White | 956 | 980 | 981 | 965 | 966 | 4848
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 43 | 30 | 38 | 33 | 36 | 180
Political Affiliation [Count of Participants; unit: Participants]
  Republican | 422 | 437 | 432 | 434 | 447 | 2172
  Democrat | 424 | 443 | 453 | 424 | 425 | 2169
  Independent | 399 | 365 | 372 | 371 | 373 | 1880
Climate Concern [Count of Participants; unit: Participants]
  Not at all | 184 | 127 | 156 | 133 | 160 | 760
  A little bit | 169 | 157 | 162 | 176 | 158 | 822
  Somewhat | 371 | 360 | 354 | 341 | 380 | 1806
  Quite a bit | 257 | 286 | 300 | 291 | 262 | 1396
  A great deal | 264 | 315 | 285 | 288 | 285 | 1437
Special Diet [Count of Participants; unit: Participants]
  No special diet | 1031 | 1010 | 1044 | 1034 | 1022 | 5141
  Vegan | 9 | 14 | 16 | 13 | 10 | 62
  Vegetarian | 29 | 21 | 25 | 24 | 28 | 127
  Pescatarian | 30 | 38 | 36 | 24 | 30 | 158
  Gluten free | 49 | 55 | 45 | 33 | 47 | 229
  Other | 97 | 107 | 91 | 101 | 108 | 504

OUTCOME MEASURES:

1. Primary Outcome: Modified Nutrient Profile Index Score
Description: The primary outcome measure will be the healthfulness of the fast-food meal selections, measured with a modified Nutrient Profile Index (NPI) score. NPI scores are based on the United Kingdom (UK) Ofcom Nutrient Profiling Model, which is used to score individual foods in the UK to determine which ones can be marketed to children. The NPI is a 0 to 100-point score for foods; scores >=64 are considered healthy. NPI awards points from nutrients to encourage (e.g., fiber, protein) and nutrients of concern (e.g., sodium, sugar) per 100 grams. The investigators will generate a modified NPI score to evaluate the healthfulness of full meals comprised of multiple food items. This measure will be determined by calculating the weighted mean NPI score of all food items selected per meal, with each item's NPI score weighted by its proportionate contribution of mass in grams to the total mass of the meal.
Time Frame: approximately 1 minute
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
Number analyzed (Participants) | 1245 | 1245 | 1257 | 1229 | 1245
score on a scale | 50.6 (0.28) | 51.3 (0.28) | 51.3 (0.28) | 50.8 (0.28) | 51.0 (0.28)

2. Secondary Outcome: Total Greenhouse Gas Emissions as Assessed by Cumulative Total Kilograms of Carbon Equivalent (kgCO2e) Per Kilogram
Description: Cumulative total kilograms of carbon equivalent (kgCO2e) per kilogram of food for all meal items.
Time Frame: approximately 1 minute
Measure: Mean (Standard Error); unit: kgCO2e/kilogram
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
Number analyzed (Participants) | 1245 | 1245 | 1257 | 1229 | 1245
kgCO2e/kilogram | 27.5 (0.97) | 23.9 (0.97) | 22.6 (0.97) | 24.6 (0.98) | 24.7 (0.97)

3. Secondary Outcome: Perceived Message Effectiveness (PME) as Assessed by the University of North Carolina (UNC) PME Scale
Description: The 3-item University of North Carolina (UNC)-PME scale measures how much the label placed beneath high climate impact menu items, discouraged consumption or evoked concern or unpleasantness about consumption of high climate impact foods. Responses to all questions will be measured on a 5-point unipolar Likert scale from 1=Not at all to 5= A great deal. Preceding the questions, participants will view the assigned label demonstrating high climate impact and the following prompt: "Considering this label, how much do you agree or disagree with the following statements." The exact text for each question is: "This label discourages me from wanting to eat foods with a high climate impact." " This label makes eating foods with a high climate impact seem unpleasant." " This label makes me concerned about eating foods with a high climate impact." The mean likert scale choice is reported. The scale choice range is between 1 and 5, with higher scores interpreted as better.
Time Frame: approximately 1 minute
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
Number analyzed (Participants) | 1245 | 1245 | 1257 | 1229 | 1245
score on a scale | 1.8 (0.05) | 2.7 (0.05) | 2.6 (0.05) | 2.5 (0.05) | 2.3 (0.05)

4. Secondary Outcome: Total Energy (Calories) Selected
Description: The total number of calories in participants' hypothetical meal orders, calculated as the sum of calories across all menu items selected. Higher values indicate more calories selected.
Time Frame: approximately 1 minute
Measure: Mean (Standard Error); unit: Calories
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
Number analyzed (Participants) | 1245 | 1245 | 1257 | 1229 | 1245
Calories | 1579.3 (17.72) | 1540.6 (25.06) | 1552.5 (25.00) | 1556.8 (25.15) | 1535.3 (25.06)

5. Secondary Outcome: Number of Participants Who Selected Sugar-sweetened Beverage
Description: Measured as a dichotomous variable (yes/no) indicating whether participants' hypothetical meal orders include a sugar-sweetened beverage.
Time Frame: approximately 1 minute
Measure: Count of Participants; unit: Participants
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
Number analyzed (Participants) | 1245 | 1245 | 1257 | 1229 | 1245
Participants | 652 | 598 | 617 | 626 | 662

ADVERSE EVENTS:
Time Frame: From enrollment to completion of survey, approximately 3 minutes.
Arm/Group | Control (QR) Labels | Warning High Climate Impact Labels | Traffic Light Labels | Climate Grade Labels | Numeric Carbon Footprint Labels
All-Cause Mortality (participants affected / at risk) | 0/1320 | 0/1339 | 0/1332 | 0/1305 | 0/1326
Serious Adverse Events (participants affected / at risk) | 0/1320 | 0/1339 | 0/1332 | 0/1305 | 0/1326
Other Adverse Events (participants affected / at risk) | 0/1320 | 0/1339 | 0/1332 | 0/1305 | 0/1326

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/78/NCT06678178/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/78/NCT06678178/SAP_001.pdf